CLINICAL TRIAL: NCT01494428
Title: A Clinical Investigation of Recombinant Human Bone Morphogenetic Protein-2 and Absorbable Collagen Sponge With Allograft Bone Dowel for Anterior Lumbar Interbody Fusion in Patients With Symptomatic Degenerative Disc Disease
Brief Title: A Pilot Study of rhBMP-2/ACS/Allograft Bone Dowel for Anterior Lumbar Interbody Fusion in Patients With Symptomatic Degenerative Disc Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-9703
Record Dates: First submitted 2011-12-12; First posted 2011-12-19 (Estimated); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Degenerative Disc Disease
Keywords: symptomatic degenerative disc disease
MeSH Terms: conditions — Intervertebral Disc Degeneration | interventions — Transplantation, Autologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- rhBMP-2/ACS (Experimental)
  Interventions: Device: rhBMP-2/ACS/allograft bone dowel
- Autogenous Bone (Active Comparator)
  Interventions: Device: Autogenous bone/allograft bone dowel

INTERVENTIONS:
Device: rhBMP-2/ACS/allograft bone dowel — The rhBMP-2/ACS will be used in conjunction with an allograft bone dowel.
  Other Names: Recombinant human bone morphogenetic protein-2
  Arms: rhBMP-2/ACS
Device: Autogenous bone/allograft bone dowel — An allograft bone dowel contains autogenous bone taken from the patient's iliac crest.
  Other Names: Autograft
  Arms: Autogenous Bone

SUMMARY:
The purpose of this pilot clinical trial is to evaluate the device design as a method of facilitating spinal fusion.

ELIGIBILITY:
Inclusion Criteria:

1. Has degenerative disc disease as noted by back pain of discogenic origin, with or without leg pain, with degeneration of the disc confirmed by patient history ( e.g.,pain [leg, back, or symptoms in the sciatic nerve distribution], function deficit and/or neurological deficit)and radiographic studies ( e.g., CT, MRl, X-Ray, etc.) to include one or more of the following:

   * instability( defined as angular motion > 5° and/or translation >= 2-4mm, based on Flex/Ext radiographs);
   * osteophyte formation;
   * decreased disc height;
   * thickening of ligamentous tissue;
   * disc degeneration or herniation; and/or
   * facet joint degeneration.
2. Has preoperative Oswestry score > 35.
3. Has no greater than Grade 1 spondylolisthesis utilizing Meyerding's Classification (Meyerding HW, 1932.).
4. Has single-level symptomatic degenerative involvement from L4 to S1.
5. Is at least 18 years of age, inclusive, at the time of surgery.
6. Has not responded to non-operative treatment (e.g., bed rest, physical therapy, medications, spinal injections, manipulation, and/or TENS) for a period of at least 6 months.
7. If female of child-bearing potential, who is not pregnant or nursing, and who agrees to use adequate contraception for 16 weeks following surgery.
8. Is willing and able to comply with the study plan and sign the Patient Informed Consent Form.

Exclusion Criteria:

1. Had previous anterior spinal fusion surgical procedure at the involved level.
2. Has a condition which requires postoperative medications that interfere with fusion, such as steroids or nonsteroidal antiinflammatory drugs (this does not include low dose aspirin for prophylactic anticoagulation).
3. Has osteopenia, osteoporosis, or osteomalacia to a degree that spinal instrumentation would be contraindicated.
4. Has presence of active malignancy.
5. Has overt or active bacterial infection, either local or systemic.
6. Is obese, i.e., weight greater than 40% over ideal for their age and height.
7. Has fever (temperature> 101° F oral) at the time of surgery.
8. Is mentally incompetent. If questionable, obtain psychiatric consult.
9. Has a Waddell Signs of Inorganic Behavior score of 3 or greater.
10. Is a prisoner.
11. Is an alcohol and/or drug abuser.
12. Is a tobacco user at the time of surgery.
13. Patient has received drugs which may interfere with bone metabolism within two weeks prior to the planned date of spinal fusion surgery (e.g., steroids or methotrexate).
14. Patient has a history of autoimmune disease (Systemic Lupus Erythematosus or Dermatomyositis).
15. Patient has a history of exposure to injectable collagen implants.
16. Patient's history includes hypersensitivity to protein pharmaceuticals (monoclonal antibodies or gamma globulins) or collagen.
17. Patient has received treatment with an investigational therapy within 28 days prior to implantation surgery or such treatment is planned during the 16 weeks following rhBMP-2/ACS implantation.
18. Patient has received any previous exposure to BMP.
19. Patient has a history of severe allergy, an allergy to bovine products, or a history of anaphylaxis.
20. Patient has history of endocrine or metabolic disorder known to affect osteogenesis (e.g., Paget's disease, renal osteodystrophy, Ehlers-Danlos syndrome, or osteogenesis imperfecta).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 1998-04; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Severity and Rate of Implant-Associated Adverse Events | 24 month
Rate of Implant Revision, Removal and Supplemental Fixation Procedures | 24 month
Incidence of Permanent Adverse Events | 24 month
Fusion | 24 month
  Fusion is defined as:
  1. Bone observed connecting with the vertebral bodies above and below either through the implants; lateral to or between the implants; or anterior/posterior to the implants.
  2. Angulation < 5°.
  3. Translation < 3mm.
  4. Absence of radiolucent lines around more than 50% of either implant.
Disc Height Measurement | 24 month
  Disc height will be measured postoperative and compared to the preoperative measurement. Maintenance or improvement in disc height will be determined a success.
Pain/Disability Status | 24 month
  The self-administered Oswestry Low Back Pain Disability Questionnaire will be used. Success will be defined as pain/disability improvement postoperatively according to the following definition: Preoperative Score - Postoperative Score >= 15
Neurological Status | 24 month
  Neurological status will be assessed preoperatively and postoperatively using a comprehensive neurological status scale.

SECONDARY OUTCOMES:
Nature and Frequency of Adverse Events Not Associated with the Implants | 24 month
Rate of Reoperation Procedures | 24 month
Hip (Donor Site) Pain Status | 24 month
Patient Satisfaction/Quality of Life Status (SF-36) | 24 month
Pain Status (Numerical Rating Scale) | 24 month
Overall Success | 24 months
  A patient will be considered an overall success if all of the following conditions are met:
  1. fusion
  2. disc height maintenance or improvement
  3. pain/disability (Oswestry) improvement
  4. maintenance or improvement in neurological status
  5. no permanent adverse event
  6. no additional surgical procedure classified as a "failure."